CLINICAL TRIAL: NCT02027272
Title: Eclampsia and Posterior Reversible Encephalopathy Syndrome (PRES): A Randomized Clinical Trial Evaluating Corticosteroid Efficacy to Augment Standard Therapy and Shorten Recovery.
Brief Title: Eclampsia and Posterior Reversible Encephalopathy Syndrome (PRES):
Acronym: PRESIDEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting, only one participant in 18 months, rarity of event
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, James Martin, Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0269
Record Dates: First submitted 2013-01-15; First posted 2014-01-06 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Eclampsia
Keywords: Eclampsia
MeSH Terms: conditions — Eclampsia | interventions — Dexamethasone; Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 12 mg, 2 doses, 12 hours apart.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo, 2 doses, 12 hours apart
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Intravenous Dexamethasone 12 mg, 2 doses, 12 hours apart
  Other Names: Potent glucocorticoid or steroid

SUMMARY:
This is a double blinded, placebo-controlled trial to determine if IV dexamethasone more quickly than placebo assists resolution of Posterior Reversible Encephalopathy Syndrome (PRES) encountered in eclamptic patients. All patients regardless of assignment to placebo or steroid will receive standard therapy to include magnesium sulfate, blood pressure medications and diuretics. We hypothesize that the addition of dexamethasone to standard therapy will accelerate CNS recovery more quickly than standard management without dexamethasone.

DETAILED DESCRIPTION:
30 eclamptic patients who do not require steroids for fetal lung maturation purposes will be randomized to placebo or steroid. This includes patients with eclampsia encountered antepartum prior to 23 weeks gestation, postpartum eclampsia, undelivered patients encountered after 33 weeks gestation who would not be candidates for fetal lung maturation steroids, or patients not eligible for repeat steroid administration in the 23-34 week gestational window. Planned enrollment in this pilot study is up to 30 patients with at least 12 in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Currently 34 weeks pregnant or within 6 weeks postpartum
2. At least 18 years of age
3. Singleton or twin gestation
4. Patient or family sign informed consent
5. Diagnosis of eclampsia
6. Able to obtain MRI scanning within 24hours of hosp admit and/or seizure

Exclusion Criteria:

1. Neither pregnant nor within first 6 weeks postpartum
2. Patient or family unable to sign informed consent
3. Less than 18 years of age
4. Triplet or higher order gestation
5. Unable to obtain MRI scanning within 24 hours of hospital admission (
6. Diagnosis of cerebral hemorrhage
7. Patient in whom MRI is contraindicated

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Martin, MD, Principal Investigator — University of Mississippi Medican Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Gender [Number; unit: participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Eclampsia and Posterior Reversible Encephalopathy Syndrome (PRES): Arandomized Clinical Trial Evaluating Corticosteroid Efficacy to Augment Standard Therapy and Shorten Recovery
Description: To learn if giving IV dexamethasone to eclamptic women with PRES will accelerate normalization of CNS function.
Time Frame: 36 months
Population: Logistic hurdles caused to stop the study after the first participant and not proceed further. No analysis was undertaken.
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No AE.
Description: No AE
Arm/Group | Dexamethasone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes